CLINICAL TRIAL: NCT05170737
Title: A First-In-Human Phase I Study in 3 Parts: Randomized, Double-blind, Placebocontrolled, Sequential Group Investigation of the Safety, Tolerability, Pharmacokinetics of AEF0217 After Oral, Single and Multiple Ascending Doses, and an Open Label, Cross-over Investigation of the Effect of Food on the Bioavailability of AEF0217 in Healthy Volunteers.
Brief Title: AEF0217 First-in-Human Phase I Study in 3 Parts (Single and Multiple Ascending Doses, and Food Effect) in Healthy Subjects.
Acronym: AEF0217-101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aelis Farma (Industry)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AEF0217-101; 2020-005201-99 (EudraCT Number)
Record Dates: First submitted 2021-12-07; First posted 2021-12-28 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Safety, Tolerability, Pharmacokinetics of AEF0217

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PART I: SINGLE ASCENDING DOSE (FIH-SAD) (Experimental): Prospective, monocenter, double-blind, randomized, placebo-controlled, subsequent-group, Phase I investigation to assess the safety, tolerability and pharmacokinetics of AEF0217 administered orally in single ascending doses.
  Interventions: Drug: AEF0217; Drug: Placebo
- PART II: MULTIPLE ASCENDING DOSES (FIH-MAD) (Experimental): Prospective, monocenter, double-blind, randomized, placebo-controlled, subsequent-groups, Phase I investigation to assess the safety, tolerability and pharmacokinetics of AEF0217 administered orally in multiple ascending doses.
  Interventions: Drug: AEF0217; Drug: Placebo
- PART III: FOOD EFFECT (FIH-FE) (Experimental): Prospective, open-label single dose, two-condition (fed versus fasting), two sequences, crossover phase I investigation to assess the effects of food on the bioavailability of AEF0217.
  Interventions: Drug: AEF0217

INTERVENTIONS:
Drug: AEF0217 — PART I: A total of 32 healthy male and female subjects will be randomized into four consecutive single ascending dose cohorts of 8 subjects. The study will have 4 different doses of AEF0217 (0.2, 0.6, 2 & 6 mg) and 1 dose of matching placebo. A given subject can be randomized only in one dose level cohort.
  PART II: A total of 24 healthy subjects will be randomized in three consecutive multiple ascending dose cohorts of 8 subjects. The study will have 3 different doses of AEF0217 (0.6, 2 & 6 mg) and 1 dose of matching placebo. Doses could be modified following the results of FIH-SAD. A given subject can be randomized only in one dose level cohort.
  PART III: A total of 12 healthy male subjects will be randomly assigned to one of two sequences in the crossover study part. All subjects will receive the same dose of AEF0117 which will be determined following the results of the FIH-SAD.
  Other Names: 3ß-benzyloxy-17α-methyl-pregn-5-en-20-one
Drug: Placebo — PART I: A total of 32 healthy male and female subjects will be randomized into four consecutive single ascending dose cohorts of 8 subjects. The study will have 4 different doses of AEF0217 (0.2, 0.6, 2 & 6 mg) and 1 dose of matching placebo. A given subject can be randomized only in one dose level cohort.
  PART II: A total of 24 healthy subjects will be randomized in three consecutive multiple ascending dose cohorts of 8 subjects. The study will have 3 different doses of AEF0217 (0.6, 2 & 6 mg) and 1 dose of matching placebo. Doses could be modified following the results of FIH-SAD. A given subject can be randomized only in one dose level cohort.
  Arms: PART I: SINGLE ASCENDING DOSE (FIH-SAD); PART II: MULTIPLE ASCENDING DOSES (FIH-MAD)

SUMMARY:
This trial is divided in 3 parts: FIH-SAD (Single Ascending Doses), FIH-MAD (Multiple Ascending Doses) and FIH-FE (Food effects). FIH-SAD will start first. The start of FIH-MAD will await the results of at least three cohorts from the FIHSAD study before initiated. The starting dose of the FIH-MAD will have been shown to be well tolerated and one dose level lower than the highest dose for which safety, tolerability and pharmacokinetic (PK) data are available. FIH-FE will be the last to start after the completion of FIH-SAD and conducted in parallel with parts of FIH-MAD.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects: As the effect of the study drug on sperm is still unknown, male subjects should refrain from donating sperm or plan a pregnancy with their partner throughout the study and until 90 days after the trial and must report immediately to the study doctor if its partner becomes pregnant during the trial and during 90 days after the trial. The male subject will have to use double-barrier contraceptive methods: male condoms and spermicide.
* Healthy female subjects of non-child-bearing potential: females may be accepted if they are documented to be surgically sterile i.e., hysterectomy, tubal ligation or post-menopausal with a negative pregnancy test (Not applicable for FIH-FE part III as it includes male only)
* Age ≥ 18 and ≤ 55 years.
* Weight ≥ 50 kg and ≤ 100 kg.
* Body mass index (BMI) ≥ 18 and ≤ 30.
* Negative serum pregnancy test (women only)
* Non-smoking.
* No history of or ongoing clinically relevant diseases or conditions.
* No clinically relevant findings in physical examination, vital signs (blood pressure, heart rate and body temperature), ECG and safety laboratory parameters that should be within normal ranges or considered as non-clinically relevant by the investigator.
* Negative covid19 PCR test within 72h before admission
* Able/willing to accept restrictions regarding diet, physical exercise, and consumption of alcohol and/or xanthine containing items when out of CRU.
* Able to read Spanish and adhere to study requirements.
* Not under any administrative or legal supervision.
* Signed informed consent prior to any study-mandated procedure.

Exclusion Criteria:

* Women of child-bearing potential
* Life-time substance use disorders (SUD) according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5).
* Recreational use of drugs of abuse within the last month prior to study drug administration.
* Positive blood or urine test for drugs of abuse or alcohol breath test prior to study drug administration.
* Life-time history of bipolar disorders, psychosis or suicidal attempts assessed by the Dual Diagnosis Screening Instrument (DDSI).
* History of anxiety or depression not completely recovered within 12 months prior to study drug administration, as assessed by the DDSI.
* Lifetime history of deliberate self-harm due to suicidal ideation or suicidal ideation prior to study drug administration, as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS).
* Clinically relevant cognitive impairment preventing the administration of the psychometric tests
* Any other clinically relevant disease or condition that in the judgment of the investigator might interfere with the subject's ability to comply with study procedures or requirements and/or bias the interpretation of the study results and/or jeopardize the subject's safety.
* Ongoing gastrointestinal diseases or history of gastrointestinal surgery affecting absorption
* Subjects with a clinically significant disease within one month prior to study drug administration.
* Any clinically relevant findings in physical examination, vital signs, ECG and safety laboratory parameters.
* Positive hepatitis or HIV test.
* Positive Covid19 PCR test within 72h before admission (Day -1) to the research facility
* Have abnormal screening values for the steroid hormones: cortisol, testosterone, estradiol and progesterone relative to their reproductive status.
* Known hypersensitivity to any drug (in particular steroids) or drug excipients.
* Use of drugs known to induce or inhibit hepatic drug metabolism within one month prior to study administration or during the study and use of citrus juice during the study.
* Any prescription or over-the-counter (OTC) product including herbal, homeopathic, vitamins, minerals and nutritional supplements and in particular any parenteral or topical product containing steroids, within 2 weeks (or more considering the elimination half-life of the product) prior to study drug administration
* Donation of blood or plasma within one month prior to study drug administration or transfusion of blood or plasma for medical/surgical reasons or intention to donate blood or plasma within one month after study drug administration.
* History of inadequate venous access and/or experience of difficulty donating blood.
* Not able/not willing to accept restrictions regarding diet, physical exercise, and consumption of alcohol and/or xanthine containing items when out of CRU.
* Subject included in a clinical study within 3 months prior to study drug administration.
* Subject already included in other parts of this study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent AEs and SAEs as assessed by vital signs | 168 hours from dosing
  Evaluation by grade intensity and by evaluating changes from the baseline in vital signs Treatment-emergent potentially clinically significant abnormalities (PSCAs) in vital signs, ECG and safety laboratory parameters from Day 1 to EOS.
  Psychopathological tests: Profile of Mood States 2nd edition questionnaire (POMS-2), Hospital Anxiety and Depression rating scale (HADS), Addiction Research Center Inventory 49 checklist (ARCI-49), Columbia-Suicide Severity Rating Scale (C-SSRS)
Incidence of treatment-emergent AEs and SAEs as assessed by ECGs | 168 hours from dosing
  Evaluation by grade intensity and by evaluating changes from the baseline in ECGs
Incidence of treatment-emergent AEs and SAEs as assessed by clinical laboratory values | 168 hours from dosing
  Evaluation by grade intensity and by evaluating changes from the baseline in clinical laboratory values from blood and urine samples.
Incidence of treatment-emergent AEs and SAEs as assessed by psychometric tests | 36 hours from dosing
  Evaluation by grade intensity and by evaluating changes from the baseline in psychometric tests (Bond and Lader VAS, ARCI, POMS) and C-SSRS test.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael de la Torre Fornel, PhD, Principal Investigator — IMIM
Locations (1):
- Hospital del Mar Medical Research Institute (IMIM) Neurosciences Research Program, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No